CLINICAL TRIAL: NCT04361266
Title: Use of Nanoscaffold Augmentation in Rotator Cuff Repair: Clinical Outcome and Ultrasound Assessment of Healing Rates and Vascularity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn
Sponsor: Joshua Szabo, MD (Other)
Collaborators: Atreon Orthopedics (Industry)
Responsible Party: Sponsor-Investigator, Joshua Szabo, MD, Clinical Instructor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19080165
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Rotator Cuff Syndrome of Shoulder and Allied Disorders
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: prospective randomized control trial
Who Masked: Investigator
Masking Description: Blinded ultrasound assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotium patch recipient (Experimental): Subjects with Rotium nano scaffold patch included in rotator cuff repair construct
  Interventions: Device: Rotium nanoscaffold
- Control (Active Comparator): Subjects undergoing non-patch augmented rotator cuff repair
  Interventions: Procedure: Control arm rotator cuff repair

INTERVENTIONS:
Device: Rotium nanoscaffold — Rotium bioabsorbable nanoscaffold placed between bone-tendon interface of rotator cuff repair construct
  Arms: Rotium patch recipient
Procedure: Control arm rotator cuff repair — Standard rotator cuff repair without Rotium
  Arms: Control

SUMMARY:
The purpose is to assess Rotium, a novel nanoscaffold, impact on healing of a repaired rotator cuff and compare to a repair without Rotium. Animal (sheep) models have shown both quicker and more organized healing when Rotium is used, but there are no studies to confirm these outcomes translate to human population.

Hypothesis: Rotium rotator cuff repairs will heal both quicker and better than traditional rotator cuff repair techniques.

DETAILED DESCRIPTION:
Patients indicated for rotator cuff repair surgery will be offered participation within the study and consented accordingly. A copy of the consent will be provided to the participant. A preoperative ultrasonographic assessment will occur by Dr. Onishi. A randomization process by computer program will determine patients who have Rotium augmented repairs, or not. The patients will not be blinded.

The surgery will be carried out by a single surgeon making all aspects uniform, except if there is or is not a Rotium patch. The Rotium patch will be implanted in accordance to standards of handling sterile implants and placed in a manner that is consistent to its FDA approval. The patch will be furnished by the institution where the surgery is being performed. Digital photography will document pertinent arthroscopic operative findings per standard of care.

Participant assessment will commence preoperatively in an outpatient clinic then continue in postoperative period, occurring at 2, 4, 6 weeks and 3, 6 and 12 month intervals. During each visit, the participants will be assessed by two clinicians: the principal investigator and a blinded ultrasonographer.

Preoperative assessment will include obtaining baseline patient reported outcomes (UCLA, Rowe, Constant, American Shoulder and Elbow Surgeons (ASES) score and SANE (Single Alpha Numeric Evaluation)scores) by paper questionnaire. A medical history will document NSAID use, cortisone injections about the shoulder, tobacco usage, narcotic medicine consumption, and pregnancy status. Due to their deleterious effects on healing, all patients will be instructed to not take NSAIDs in the first 6 weeks postoperative. Noncompliance will be noted, but not disqualify the participant from study. Smoking cessation will be strongly encouraged. A shoulder physical examination will be performed; specifically range of motion assessment in multiple planes (frontal flexion, internal and external rotation at 90 degrees of abduction and at side), rotator cuff muscle strength testing with the scapula stabilized, scapula posture observed, and provocative tests for impingement syndrome. Medical records will be reviewed. This evaluation will be performed by the principal investigator and will take 45-60 minutes. The participant will undergo a separate diagnostic ultrasonographic assessment of the rotator cuff tendons by blinded ultrasonographer. This will take 15-30 minutes.

Aftercare of each population will be identical and will include a 6-week period of sling immobilization, brief perioperative narcotic medicine, and physical therapy. Physical therapy protocols will be identical. The participants will be treated by a variety of physical therapists. All physical therapy will occur out of the home at a PT clinic. Additional home exercises will be furnished and will be independently performed by the participants.

Specifically, at the 2-week postoperative visit a history will be obtained to quantify narcotic usage, NSAID usage, VAS pain score, and assess for any complications. The surgical site and sling will be inspected, passive range of motion of the shoulder assessed (frontal flexion and external rotation at the side), and the examine will exclude any complications. Physical therapy for shoulder passive range of motion and periscapular strengthening will be prescribed, home exercise sheet provided, and the abduction portion of the sling will be discontinued. Shoulder radiographs will be performed. This visit will take 15-30 minutes. In addition and separate to this,blinded ultrasonographer will perform ultrasound assessment of the repaired rotator cuff. Vascularity using superb microvascular imaging and standard ultrasound techniques will assess vascularity and rotator cuff repair integrity. If possible, elastography will be performed. These images will be stored in de-identified manner within University of Pittsburgh HIPPA-compliant cloud. This will take 15-30 minutes and may be done at a separate time.

At the 4-week postoperative visit a history will be obtained to quantify narcotic usage, NSAID usage, pain score, and assess for any complications. The surgical site and sling will be inspected, passive range of motion of the shoulder (frontal flexion and external rotation at the side) assessed, and the examine will exclude any complications. The prior physical therapy and home exercises will be continued. This visit will take 15-30 minutes. In addition and separate to this, blinded ultrasonographer will perform ultrasound assessment of the repaired rotator cuff. This will take 15-30 minutes and may be done at a separate time.

At the 6-week postoperative visit a history will be obtained to quantify narcotic usage, NSAID usage, pain score, and assess for any complications. The surgical site and sling will be inspected, passive range of motion of the shoulder (frontal flexion, internal and external rotation at 90 degrees of abduction and at side) assessed, and the examine will exclude any complications. The sling will be discontinued and new physical therapy and home exercises will be provided; therapy will include shoulder passive range of motion and periscapular strengthening and include rotator cuff strengthening progressing from isometric to concentric then to eccentric with the pace being determined by a physical therapist, but done in a pain free manner. Additionally, patient reported outcomes (UCLA, Rowe, Constant, ASES and SANE scores) will be collected. This visit will take 30-45 minutes. In addition and separate to this, blinded ultrasonographer will perform ultrasound assessment of the repaired rotator cuff. This will take 15-30 minutes and may be done at a separate time.

At the 3-, 6- and 12-month postoperative visits a history will be obtained to assess shoulder functionality/limitations, quantify NSAID usage, pain score, and assess for any complications. The examination will be similar to the 6-week evaluation, except rotator cuff specific strength will be assessed similar to the preoperative testing. Necessity of ongoing physical therapy will be considered and ordered appropriately. Home exercises will be continued. These visits will take 30-45 minutes. In addition and separate to this, blinded ultrasonographer will perform ultrasound assessment of the repaired rotator cuff. This will take 15-30 minutes and may be done at a separate time.

ELIGIBILITY:
Inclusion Criteria:

* -symptomatic supraspinatus or supraspinatus and infraspinatus tear that can be repaired to the greater tuberosity in an anatomical manner using a dual layer repair technique.
* also included will be patients that have concomitant pathology addressed at time of surgery, specifically pathologies of the biceps tendon (tenodesis or tenotomy), arthrosis of the acromioclavicular joint (distal clavicle resection), or labral tearing (debridement or repair)
* included age range of subjects will be from 18-80 years old

Exclusion Criteria:

* diabetes, cancer or medical states that may impair healing, such as organ transplantation or systemic inflammatory process treated with immune modulating drugs (chemotherapy, immunosuppression drugs)
* prior surgery to the ipsilateral rotator cuff tendon
* need of soft tissue releases to accomplish an anatomic repair, partial repairs and/or concomitant subscapularis repair
* significant glenohumeral arthritis
* active or ongoing infection
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff integrity baseline/preoperative | preoperative
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 2 weeks | postoperative at 2 weeks
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 4 weeks | postoperative at 4 weeks
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 6 weeks | postoperative at 6 weeks
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 3 months | postoperative 3 months
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 6 months | postoperative at 6 months
  ultrasound assessment of rotator cuff
Rotator cuff repair integrity @ 12 months | postoperative at 12 months
  ultrasound assessment of rotator cuff
Postoperative rotator cuff vascularity during healing | postoperative at 2 weeks
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)
Postoperative rotator cuff vascularity during healing | postoperative at 4 weeks
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)
Postoperative rotator cuff vascularity during healing | postoperative at 6 weeks
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)
Postoperative rotator cuff vascularity during healing | postoperative at 3 months
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)
Postoperative rotator cuff vascularity during healing | postoperative at 6 months
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)
Postoperative rotator cuff vascularity during healing | postoperative at 12 months
  ultrasound assessment of rotator cuff at repair site using superb microvascular imaging (SMI)

SECONDARY OUTCOMES:
University California Los Angeles Shoulder score | preoperative and postoperative at 6 weeks and 3,6,12 months postoperative
  Outcome score
Rowe score | preoperative and postoperative at 6 weeks and 3,6,12 months postoperative
  Outcome score
Constant score | preoperative and postoperative at 6 weeks and 3,6,12 months postoperative
  Outcome score
American shoulder and elbow surgeons score | preoperative and postoperative at 6 weeks and 3,6,12 months postoperative
  Outcome score
SANE score | preoperative and postoperative at 2,4, 6 weeks and 3,6,12 months postoperative
  Outcome score

OTHER OUTCOMES:
NSAID usage | postoperative period @ 2,4, 6 weeks and 3, 6, 12 months
  total dosage of NSAIDs
Cortisone injections about the shoulder | preoperative period
  Include total number and timeframe relative to surgical date
Tobacco usage | preoperative and postoperative periods @ 2,4, 6 weeks and 3, 6, 12 months
  Daily consumption
Narcotic consumption | postoperative period @ 2,4, 6 weeks and 3, 6, 12 months
  total dosage of narcotic medicine

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time.